CLINICAL TRIAL: NCT05775432
Title: Prognosis of Heart Transplanted Patients With Heart Failure (RE-START): a National Multi-center, Retrospective-prospective, Cohort Study
Brief Title: Prognosis of Heart Transplanted Patients With Heart Failure
Acronym: RE-START
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-391
Record Dates: First submitted 2023-02-14; First posted 2023-03-20 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure
Keywords: Heart transplantation; Heart failure; Prognosis
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood, urine, feces.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heart transplantation group: Patients with heart failure of different etiologies undergoing heart transplant.
- Control group: Individuals whose hearts are donated.

SUMMARY:
Heart transplantation is the most effective treatment for end-stage heart failure, advanced cardiomyopathy, and complex congenital heart disease with severe heart failure or hypoxia. Several clinical studies have shown significant differences in the prognosis of heart transplantation patients with different etiologies, and post-transplantation complications are an important factor affecting patient survival, and there is still a lack of overall prognostic stratification and extensive clinical studies on risk factors after heart transplantation. Therefore, this study is intended to include patients who underwent heart transplantation for different etiologies of heart failure, collect clinical data and biological samples from patients, and use various techniques to deeply interpret the risk factors affecting the prognosis of heart transplantation patients and construct a prognostic prediction model to provide specific and individualized treatment ideas and theoretical basis for improving the survival rate of patients after heart transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end-stage heart failure presented to our hospital who are evaluated by clinicians and ethically approved for heart transplantation
* Individuals whose hearts are donated

Exclusion Criteria:

* Patients refuse to sign informed consent form

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with end-stage heart failure presented to our hospital who are evaluated by clinicians and ethically approved for heart transplantation are enrolled into heart transplantation group. Individuals whose hearts are donated are enrolled into control group.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-04-23 (Actual); Primary Completion 2042-12-31 (Estimated); Study Completion 2042-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the incidence of all-cause death | In-hospital (an average of 1 month), 1, 2, 3, 5, 10, 15 and 20 years after heart transplantation.
  Death from any cause in patients after heart transplantation, will be assessed from medical records.

SECONDARY OUTCOMES:
Use of advanced life support (ALS) | In-hospital (an average of 1 month)
  Duration of ALS after heart transplantation, will be assessed from medical records.
Incidence of postoperative complications | In-hospital (an average of 1 month)
  Postoperative complications after heart transplantation will be assessed from medical records.
ICU admission time | In-hospital (an average of 1 month)
  ICU admission time after heart transplantation, will be assessed from medical records.
Change of cardiac function index | In-hospital (an average of 1 month).
  Cardiac functional index after heart transplantation will be assessed by transthoracic echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Li, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; Yang Yan, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided